CLINICAL TRIAL: NCT00174512
Title: A Methodological Open-Label Cross-Over Controlled Study To Assess The Effect Of Drugs On Ventricular Repolarisation and QT Interval At Fixed Heart Rate Under Autonomic Blockade
Brief Title: A Methodological Open Label Cross-Over Controlled Study To Assess The Effect Of Drugs On Ventricular Repolarization and QT Interval At Fixed Heart Rate Under Autonomic Blockade
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: A9001226
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-11-08 (Estimated); Status verified 2006-11

CONDITIONS: Patients With Pace Makers But no Evidence of Ischemic Heart Disease
MeSH Terms: interventions — Moxifloxacin

INTERVENTIONS:
Drug: GTN
Drug: Moxifloxacin

SUMMARY:
To assess the effects of GTN on QT and QTc in subjects with And without atrial pacing. This will be done with and without autonomic blockade at two different pacing rates. Moxifloxacin effect on QT and QTc will also be assessed in atrially paced patients at two different pacing rates with and without autonomic blockade

ELIGIBILITY:
Inclusion Criteria:

* Patients with pace-makers but otherwise normal ventricular function

Exclusion Criteria:

* Nitrates, beta blockers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2005-03; Study Completion 2006-06

PRIMARY OUTCOMES:
QT and QTc changes at two different pacing rates in atrially paced patients

SECONDARY OUTCOMES:
Change in QT and QTcF before and after Moxifloxacin with and without autonomic blockade at each pacing rate Change in QT and QTcF before and after autonomic blockade at each pacing rate

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Pfizer Investigational Site, Bruxelles (Brussels), Belgium
- United Kingdom (5):
  - Pfizer Investigational Site, Glasgow, Scotland
  - Pfizer Investigational Site, Leicester
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001226&StudyName=A+Methodological+Open+Label+Cross%2DOver+Controlled+Study+To+Assess+The+Effect+Of+Drugs+On+Ventricular+Repolarization+and+QT+Interval+At+Fixed+Heart+Rate+Under+Autonomic+Bloc